CLINICAL TRIAL: NCT01294670
Title: A Phase I/II Clinical Study of Vorinostat in Combination With Etoposide in Pediatric Patients < 21 Years at Diagnosis With Refractory Solid Tumors
Brief Title: Clinical Study of Vorinostat in Combination With Etoposide in Pediatric Patients < 21 Years at Diagnosis With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Phoenix Children's Hospital (Other); Milton S. Hershey Medical Center (Other); Johns Hopkins University (Other); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other); Children's Hospital Colorado (Other); University of Florida (Other); Alberta Children's Hospital (Other); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other); Children's Mercy Hospital Kansas City (Other); Johns Hopkins All Children's Hospital (Other); Arnold Palmer Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-096
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumors; Relapsed/Refractory Sarcomas
Keywords: ETOPOSIDE (VP-16); SAHA (SUBEROYLANILIDE HYDROXAMIC ACID) (Vorinostat); Pediatric; 10-096; POETIC; phase II component: the population will be restricted to relapsed/refractory sarcomas.
MeSH Terms: conditions — Sarcoma | interventions — Vorinostat; Etoposide

ARMS (1):
- Vorinostat and Etoposide (Experimental): This is a multi-center, open label, phase I/II trial of escalating doses of vorinostat in combination with etoposide.
  Interventions: Drug: Vorinostat and Etoposide

INTERVENTIONS:
Drug: Vorinostat and Etoposide — Patients will be assessed in 3-week cycles. Escalating doses of vorinostat will be administered orally on a daily x 4 schedule in combination with a fixed dose of etoposide. Etoposide will be administered intravenously daily x 3 days. Cohorts of 3-6 patients will be treated with vorinostat and etoposide. In the phase II component, patients will be treated at the RP2D established in the Phase I component of the study, which was found to be 270 mg/m2/dose of Vorinostat and 100 mg/m2/dose of Etoposide.

SUMMARY:
The purpose of this study is to find out how safe and effective treatment with a new combination of drugs, vorinostat and etoposide, is in treating cancer. The medication etoposide is a standard medication used in the treatment of cancer in children. Vorinostat is an experimental drug which targets a protein(s) that control the way cancer cells grow and divide. Vorinostat is approved by the FDA in adults with certain cancers but not approved yet in children.

There are two parts to this study. In the first part of this study, the phase I portion, a safe dose of the combination, vorinostat and etoposide. The goal of second part of this study, the phase II portion, is to see how effective the combination of vorinostat and etoposide is in treating cancer.

ELIGIBILITY:
Inclusion Criteria:

* Phase I Component: Histologic confirmation of relapsed/refractory solid tumors, including tumors of the central nervous system that have failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist. Patients with diffuse pontine glioma are not required to have histologic confirmation of disease, and are eligible with radiologic confirmation. Phase II Component: the population will be restricted to relapsed/refractory sarcomas
* Patient must be between 4-21 years of age at the time of study enrollment. Efforts will be made to enroll patients <13 years of age so that adequate information about the biologic effects of this agent in younger patients can be obtained.
* Patient must have Karnofsky > or = to 60% for patients >10 years of age; Lansky Play Scale > or = to to 60 for children < or = to 10 years of age
* Patient must have a life expectancy of > 8 weeks.
* There is no limit to the number of prior treatment regimens provided that performance status and life expectancy meet the criteria above.
* Absolute neutrophil count (ANC) ≥ 1000 / mcL
* Platelets ≥100,000 / mcL (transfusion not permitted)
* Hemoglobin ≥ 9 g/dL qualifications (transfusion permitted)
* Coagulation Prothrombin Time or INR ≤ 1.5x upper limit of normal (ULN)
* Serum creatinine ≤ 1.5x upper limit of normal (ULN) OR calculated creatinine clearance ≥ 60 mL/min for patients with creatinine levels > 1.5x institutional ULN. or calculated creatinine clearance Creatinine clearance should be calculated per institutional standard.
* Serum total bilirubin ≤ 1.5 x ULN Patient's who don't meet this criteria must have a Direct bilirubin ≤ 1.5 x ULN
* AST (SGOT) and ALT (SGPT) Alkaline Phosphatase (liver fraction)

  ≤ 2.5 x ULN. If AST or ALT is > 2.5 x ULN, then the liver fraction of Alkaline Phosphatase should be ≤ 2.5 x ULN
* Phase I component: Patients may have measurable or non-measurable disease. Phase II component: Patients may only have measurable disease.
* Patient must have no persistent toxicities from prior therapy > or = to Grade 2 with the exception of hematologic indices (i.e. hemoglobin, WBC, ANC, ALC).
* For females of childbearing potential, a negative serum pregnancy test must be documented within 72 hours of receiving the first dose of vorinostat.
* Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent.
* Female patients of childbearing potential must be willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study, starting with visit 1.
* Male patients must agree to use an adequate method of contraception for the duration of the study.
* Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: At least 2 weeks must have elapsed since the administration of previous therapy. Six weeks must have elapsed since administration of nitrosoureas or mitomycin C. Seven days must have elapsed since the administration of G-CSF and/or GM-CSF.
* Biologic agents: At least 14 days must have elapsed since the completion of therapy with a biologic agent such as a monoclonal antibody. Seven days must have elapsed since the last dose of retinoids.
* Radiation therapy (XRT): > or = to 2 weeks must have elapsed for local XRT (small port); > or = to 6 months must have elapsed if prior radiation to > or = to 50% of the pelvis or if other substantial bone marrow irradiation, including total body irradiation.
* Patient must be able to swallow capsules.
* Patient must have an available archival/pre-treatment block or fresh tumor biopsy for molecular profiling to be performed.

Exclusion Criteria:

* A patient meeting any of the following criteria is not eligible to participate in this study:
* Patients currently participating or has participated in a study with an investigational compound or device within 4 weeks of initial dosing with study drugs.
* Patients with a prior history of treatment with HDAC inhibitors ( e.g. SNDX-275/entinostat, LAQ-824, LBH589, PXD-101/belinostat, etc). Patients who have received Valproic acid will be excluded from this study.
* Patients with non CNS primary tumors who have known brain metastases or symptomatic CNS disease (e.g. cranial nerve abnormalities) without cytologic abnormality in the CSF should be excluded from this clinical trial because of their poor prognosis and known propensity for the development of progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with metastatic CNS tumors will not be excluded from enrollment on this study in the phase I component only.
* Patients who have undergone prior autologous stem cell transplantation or allogeneic transplantation.
* Uncontrolled intercurrent illness or circumstances that could limit compliance with the study requirements including, but not limited to: ongoing or active bacterial or fungal infection, acute or chronic graft versus host disease, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations.
* Patients who are pregnant or breastfeeding, or expecting to conceive within the projected duration of the study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, lactating patients will be excluded from this study.
* Patients known to be Human Immunodeficiency Virus (HIV)-positive.
* Patients with known hypersensitivity to the components of the study drugs or their analogs.
* Patients with symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
* Patients who are at the time of signing informed consent, a regular user of any illicit drugs, substance abuser or who have a recent history of drug or alcohol abuse.
* Patients with a known history of Hepatitis B or C.
* Patients who have a history of gastrointestinal surgery or other procedures that might in the opinion of the investigator, interfere with the absorption or swallowing of the study drug.
* Patients who are unable to take or tolerate oral medications on a continuous basis.
* Patients with a history of a prior malignancy who have undergone potentially curative therapy with no evidence of that disease for five years or patients, who are deemed low risk for recurrence by his/her treating physician are permitted to enroll.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (10):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - Arnold Palmer Hospital for Children/MD Anderson Cancer Center Orlando, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - John Hopkins Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas
- Alberta Children'S Hospital, Calgary, Alberta, Canada

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 100 mg/m2 Etoposide, 125 mg/m2 Vorinostat + Data Migration
- Dose Level 2: 100 mg/m2 Etoposide, 160 mg/m2 Vorinostat + Data Migration
- Dose Level 3: 100 mg/m2 Etoposide, 210 mg/m2 Vorinostat + Data Migration
- Dose Level 4: 100 mg/m2 Etoposide, 270 mg/m2 Vorinostat + Data Migration
- Phase II: Vorinostat 270 mg/m2; Etoposide 100 mg/m2 + Data Migration
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II
Started | 7 | 3 | 3 | 9 | 5
Completed | 6 | 3 | 3 | 9 | 5
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Not treated | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II Dose: Vorinostat 270 mg/m2; Etoposide 100 mg/m2 + Data Migration
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose | Total
Number analyzed (Participants) | 7 | 3 | 3 | 9 | 5 | 27
Age, Continuous [Median (Full Range); unit: years] | 11 [6 to 17] | 12 [5 to 17] | 11.7 [4 to 16] | 10.2 [4 to 20] | 13.6 [13 to 15] | 13 [4 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 4 | 3 | 14
  Male | 4 | 2 | 0 | 5 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 7 | 3 | 2 | 8 | 3 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 1 | 0 | 5
  White | 4 | 2 | 2 | 8 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 3 | 3 | 9 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: To Establish the Dose Limiting Toxicity (DLT)
Description: of the novel combination vorinostat and etoposide in pediatric patients with refractory solid tumors including tumors of the central nervous system. The Toxicity will be evaluated according to NCI CTCAE Version 4.0.
Time Frame: Patients will be assessed in 3-week cycles.
Population: Data were not collected
Groups:
- Dose Level 1: 100 mg/m2 Etoposide, 125 mg/m2 Vorinostat (n=7)
- Dose Level 2: 100 mg/m2 Etoposide, 160 mg/m2 Vorinostat (n=3)
- Dose Level 3: 100 mg/m2 Etoposide, 210 mg/m2 Vorinostat (n=3)
- Dose Level 4: 100 mg/m2 Etoposide, 270 mg/m2 Vorinostat (n=9)
- Phase II Dose: Vorinostat 270 mg/m2; Etoposide 100 mg/m2 (n=5)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: To Establish the Maximum Tolerated Dose (MTD)
Description: of the novel combination vorinostat and etoposide in pediatric patients with refractory solid tumors including tumors of the central nervous system.
Time Frame: 1 year
Population: Data were not collected
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: To Establish the Efficacy (CR (Complete Response) + PR (Partial Response) Rate)
Description: of the novel combination vorinostat and etoposide in pediatric patients with relapsed/refractory sarcoma. Evaluation for response will be determined by Revised RECIST guideline
Time Frame: 1 year
Population: Data were not collected
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: To Evaluate the Efficacy (CR (Complete Response) + PR (Partial Response) Rate)
Description: of the novel combination vorinostat and etoposide in pediatric patients enrolled in the phase I component of the study. Evaluation for response will be determined by Revised RECIST guideline.
Time Frame: 1 year
Population: Data were not collected
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: To Evaluate the Biologic Effects Using Histone Acetylation, Gene Expression Profiling, and Histone Phosphorylation Profiling.
Description: of the novel combination of vorinostat and etoposide in pediatric patients with refractory solid tumors including central nervous system tumors
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II Dose
All-Cause Mortality (participants affected / at risk) | 5/7 | 2/3 | 1/3 | 4/9 | 3/5
Serious Adverse Events (participants affected / at risk) | 3/7 | 3/3 | 1/3 | 3/9 | 4/5
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 3/3 | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=9) | Phase II Dose (N=5)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Death NOS (General disorders) | 1 | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 2 | 2
Platelet count decreased (Investigations) | 2 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=9) | Phase II Dose (N=5)
White blood cell decreased (Investigations) | 7 | 1 | 2 | 5 | 3
Neutrophil count decreased (Investigations) | 7 | 0 | 3 | 6 | 3
Platelet count decreased (Investigations) | 6 | 0 | 1 | 4 | 2
Anemia (Blood and lymphatic system disorders) | 5 | 0 | 2 | 2 | 3
Fatigue (General disorders) | 1 | 1 | 1 | 2 | 1
Lymphocyte count decreased (Investigations) | 5 | 1 | 2 | 5 | 5
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2 | 0
Fever (General disorders) | 1 | 1 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Abducens nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 0 | 1 | 1
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Death NOS (General disorders) | 1 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT01294670/Prot_SAP_000.pdf